CLINICAL TRIAL: NCT04560231
Title: Is Remdesivir a Possible Therapeutic Option for SARS-CoV-2 : An Interventional Study
Brief Title: Remdesivir in COVID-19 Lahore General Hospital
Acronym: RC19LGH
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. M.Irfan Malik, Associate Professor of Pulmonology / Focal Person COVID-19, Lahore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH003
Record Dates: First submitted 2020-07-11; First posted 2020-09-23 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV Infection
Keywords: COVID-19; Remdesivir
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: Qausi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group intervene with Remdesivir (Experimental): Review effect of Remdesivir as clinical trial among hospitalized patients with COVID-19 infection. 200 mg I/v Remdesivir will be given to moderate disease patients of COVID-19. It will be loading dose then 100 mg I/V dose will be given for 5 days. Customized decision for Remdesivir dosage will be made by attending infectious diseases physician, comfort with usage, bacterial co-infection and duration of Ventilation and dose will be extended up to 10 days according to clinical condition of the patients.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — 200 mg I/v Remdesivir will be given to moderate disease patients of COVID-19. It will be loading dose then 100 mg I/V dose will be given for 5 days. Customized decision for Remdesivir dosage will be made by attending infectious diseases physician, comfort with usage, bacterial co-infection and duration of Ventilation and dose will be extended up to 10 days according to clinical condition of the patients.
  Other Names: Remidia

SUMMARY:
Remdesivir is a monophosphoramidate prodrug of an adenosine analogue and it has a broad-spectrum antiviral activity against paramyxoviruses, falviviruses and coronaviruses. It showed in vitro activity on human airway epithelial cells against SARS-CoV-2. It is an investigational drug and granted an Emergency Use Authorization by Food and Drug Administration FDA, so it is under clinical trial.

The potent mechanism of action of this drug is still unclear but it effects through several processes. It can interfere with nsp12 polymerase even when exoribonuclease proofreading is intact. It can also produce nucleoside triphosphate NTP that acts pharmacologically active alternate substrate of RNA-chain terminator, as a result NTP can constrain active triphosphates into viral RNA of coronaviruses. There is evidence of high genetic barrier to develop resistance against Remdesivir in coronavirus as a result of which is maintains its effectiveness in antiviral therapies against these viruses. Effectiveness of Remdesivir has been reported against different groups of coronaviruses including Alphacoronavirus NL63 and several SARS/MERS-CoV coronaviruses.

DETAILED DESCRIPTION:
This is interventional single-center study, that will be done at Lahore General Hospital in which 95 beds are allocated for COVID-19 patients including ICUs and HDUs. Ethical approval will be obtained from research ethical committee of Lahore General hospital, Lahore. Informed consent will be obtained from all patients who will agree to publish their data in this research. Patient's privacy protection will be obeyed with the Helsinki Declaration.

The aim of this study is to evaluate clinical effectiveness of this investigational drug, started a clinical trial of this drug on laboratory-confirmed COVID-19 patients at a tertiary care hospital of Lahore, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All patients of all ages, males, and females who will be diagnosed COVID-19 positive by RT-PCR with moderate illness.
* Patients having classical radiological lesions of COVID-19 on X-ray chest or HRCT chest.
* Respiratory rate > 22/ min and >50% of radiological involvement of lung with typical lesions.
* FiO2 remain static or improving along with > 30% deranged ≥ 2 biochemical markers CRP > 20 mg/l, LDH > 600 U/L, D.Dimer > 0.5mg/l or 500 ng/ml, Serum Ferritin < 500 ng/ml or mcg/l will be included in clinical trial.

Exclusion Criteria:

* Patients on Invasive mechanical ventilation (IMV).
* Patients with respiratory rate < 20/mins and whose laboratory findings will not be deranged > 20%.
* Presences of chronic renal failure > 4 stage, GFR < 30ml/min/1.73m2.
* ALT/AST > 5 times than normal values.
* Pregnant women.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response after administration | 10 days
  Clinical improvement of COVID-19 patients by Remdesivir.

SECONDARY OUTCOMES:
Clinical response to treatment | 15 days
  Overall survival of COVID-19 patients after drug administration.
Duration of hospitalization | 15 days
  Number of days of hospital admission either in ICU or HDUs till date of discharge
Supplemental Oxygen Requirement from Baseline | 15 days
  Duration of increased supplemental oxygen requirement from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Malik, FCPS, Study Director — Post-Graduate Medical Institute, Lahore General Hospital, Lahore Pakistan
Locations (1):
- Muhammad Irfan Malik, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584
- [Background] Davies M, Osborne V, Lane S, Roy D, Dhanda S, Evans A, Shakir S. Remdesivir in Treatment of COVID-19: A Systematic Benefit-Risk Assessment. Drug Saf. 2020 Jul;43(7):645-656. doi: 10.1007/s40264-020-00952-1. PMID 32468196
- [Background] Li Z, Wang X, Cao D, Sun R, Li C, Li G. Rapid review for the anti-coronavirus effect of remdesivir. Drug Discov Ther. 2020;14(2):73-76. doi: 10.5582/ddt.2020.01015. PMID 32378648